CLINICAL TRIAL: NCT06115200
Title: Norwegian Adult Mental Health Registry
Acronym: NAMHR
Status: Not yet recruiting | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: NAMHR001
Record Dates: First submitted 2023-07-03; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-05

CONDITIONS: Depression; Schizophrenia; Bipolar Disorder; Eating Disorders; Anxiety Disorders; Ptsd; Personality Disorders; Adhd
Keywords: database; epidemiology; mental health register
MeSH Terms: conditions — Depression; Schizophrenia; Bipolar Disorder; Feeding and Eating Disorders; Anxiety Disorders; Stress Disorders, Post-Traumatic; Personality Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
"The Norwegian Adult Mental Health Registry" (NAMHR) is a medical quality register collecting and systematizing data on patients and their treatment in specialist mental health care for adults in Norway. The main purpose is to create a documentation basis for quality assurance, evaluation, and improvement of assessment and treatment for patients who are offered treatment for mental disorders in the specialist health service. The register uses automatic data capture from various existing data sources. New patients are automatically included, but given the opportunity for reservations from the register without affecting their services and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Residents in Norway aged 18 years or older assessed and granted right to treatment in specialized mental in- and out-patient settings

Exclusion Criteria:

* Persons who have reserved themselves against participation
* Persons already included in more specialized register for mental disorder and/or treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents in Norway aged 18 years or older and granted right to treatment in mental specialized in- and out-patient settings (approximately 150.000 participants)
Sampling Method: Non-Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcome Measures (PROMs) | Baseline defined as: From start of treatment date (inclusion in the register) until the date of first documented assessment or date of discharge from any cause, whichever came first, assessed up to 24 months
  Percentage of subjects that experienced change in PROMs
Patient Reported Outcome Measures (PROMs) | Discharge defined as: date of discharge from any cause, assessed up to 60 months
  Percentage of subjects that experienced change in PROMs
Patient Reported Outcome Measures (PROMs) | Six months after discharge
  Percentage of subjects that experienced change in PROMs
Drug name and dosage from electronic medication management solutions | Baseline defined as: From start of treatment date (inclusion in the register) until the date of first documented assessment or date of discharge from any cause, whichever came first, assessed up to 24 months
  Frequency of psychotropic generic drug name and dosage
Drug name and dosage from electronic medication management solutions | Discharge defined as: date of discharge from any cause, assessed up to 60 months
  Frequency of psychotropic generic drug name and dosage
Drug name and dosage from electronic medication management solutions | Six months after discharge from any cause, assessed up to 12 months
  Frequency of psychotropic generic drug name and dosage
Rate of overweight defined as BMI > 25 (body mass index) | Baseline defined as: From start of treatment date (inclusion in the register) until the date of first documented assessment or date of discharge from any cause, whichever came first, assessed up to 24 months
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters.
Rate of overweight defined as BMI > 25 (body mass index) | Discharge defined as: date of discharge from any cause, assessed up to 60 months
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters.
Level of glycated haemoglobin (HbA1c) | Baseline defined as: From start of treatment date (inclusion in the register) until the date of first documented assessment or date of discharge from any cause, whichever came first, assessed up to 24 months
  Glycated hemoglobin is a form of hemoglobin chemically linked to sugar.
Level of glycated haemoglobin (HbA1c) | Discharge defined as: date of discharge from any cause, assessed up to 60 months
  Glycated hemoglobin is a form of hemoglobin chemically linked to sugar.
Level of blood pressure, both systolic and diastolic levels | Baseline defined as: From start of treatment date (inclusion in the register) until the date of first documented assessment or date of discharge from any cause, whichever came first, assessed up to 24 months
  Blood pressure varies between systolic and diastolic pressures after each heartbeat. Systolic pressure is peak (maximum) pressure in the arteries. Diastolic pressure is the lowest (minimum) pressure in the arteries.
Level of blood pressure, both systolic and diastolic levels | Discharge defined as: date of discharge from any cause, assessed up to 60 months
  Blood pressure varies between systolic and diastolic pressures after each heartbeat. Systolic pressure is peak (maximum) pressure in the arteries. Diastolic pressure is the lowest (minimum) pressure in the arteries.
Bloodlevels of total cholesterol, LDL, HDL and Triglycerides | Baseline defined as: From start of treatment date (inclusion in the register) until the date of first documented assessment or date of discharge from any cause, whichever came first, assessed up to 24 months
  A lipid profile (lipid panel) is a set blood tests used to find abnormalities in blood lipids. The present panel will include: total cholesterol, LDL, HDL and Triglycerides.
Bloodlevels of total cholesterol, LDL, HDL and Triglycerides | Discharge defined as: date of discharge from any cause, assessed up to 60 months
  A lipid profile (lipid panel) is a set blood tests used to find abnormalities in blood lipids. The present panel will include: total cholesterol, LDL, HDL and Triglycerides.
Frequency of ICD-10 or ICD-11 diagnosis F00-F99 | Baseline defined as: From start of treatment date (inclusion in the register) until the date of first documented assessment or date of discharge from any cause, whichever came first, assessed up to 24 months
  International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD-10) or ISD-11: Chapter V: Mental and behavioural disorders (F00-F99)
Frequency of ICD-10 or ICD-11 diagnosis F00-F99 | Discharge defined as: date of discharge from any cause, assessed up to 60 months
  International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD-10) or ISD-11: Chapter V: Mental and behavioural disorders (F00-F99)Revision (ICD-10) WHO: Chapter V: Mental and behavioural disorders (F00-F99)

CONTACTS AND LOCATIONS:
Overall Officials: Inge Joa, PhD, Principal Investigator — Stavanger University hospital, Stavanger, Norway